CLINICAL TRIAL: NCT04838301
Title: Safety and Efficacy of Allopregnanolone (Allo) as a Regenerative Therapeutic for Alzheimer's Disease: Multicenter, Double-Blind, Randomized, Placebo-Controlled, Phase 2 Clinical Trial
Brief Title: Allopregnanolone Regenerative Therapeutic for Mild Alzheimer's Disease
Acronym: REGEN-BRAIN©
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Syneos Health (Other); University of Southern California (Other); ADM Diagnostics (Unknown)
Responsible Party: Principal Investigator, Roberta Brinton, Director, Center for Innovation in Brain Science; Professor, Departments of Pharmacology and Neurology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Allo-20-001; R01AG063826 (NIH)
Record Dates: First submitted 2021-03-25; First posted 2021-04-09 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Dementia; Late Onset Alzheimer Disease; Neurodegenerative Diseases
Keywords: Mild Alzheimer Disease; Regenerative Therapeutic; APOE ε4; Neurogenesis; Allopregnanolone
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases | interventions — Pregnanolone

STUDY DESIGN:
Intervention Model Description: Participants are assigned to the active intervention or placebo in parallel for 12 months. After 12 months, all participants in the placebo group will be crossed-over to receive Allo for the remainder of the study (6 month open-label phase).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After 12 months participants and study personnel will be aware of the open label phase, but initial randomization will remain blind during the entire length of the study (placebo-controlled and open-label periods); that is, all participants and study personnel are blinded to each participant's randomization to initial treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allo group (Experimental): Allopregnanolone 4mg IV 30-minute infusion once per week for 12 months.
  Interventions: Drug: Allopregnanolone
- Control group (Placebo Comparator): Placebo (normal saline) IV 30-minute infusion once per week for 12 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Allopregnanolone — Allopregnanolone 4mg IV via 30-minute infusion, once per week.
  Other Names: Allo
  Arms: Allo group
Other: Placebo — Normal saline solution IV via 30-minute infusion, once per week
  Arms: Control group

SUMMARY:
A phase 2, double-blind, randomized, placebo-controlled clinical trial to evaluate the safety and efficacy of Allopregnanolone as a regenerative therapeutic for Alzheimer's disease.

DETAILED DESCRIPTION:
This is a proof-of-concept phase 2 clinical trial to investigate the long-term safety and efficacy of Allo to function as a regenerative therapeutic to restore structural integrity and cognitive function of the brain in participants with mild Alzheimer's disease (AD) dementia. Study participants will be male and female, APOE ε4 positive diagnosed with probable AD, Mini-Mental State Exam (MMSE) 20 to 26, ages 55 to 80 years old.

After a 2-4-week screening period, participants will be randomized to 4 mg Allo (administered intravenously over 30 minutes, once per week, in clinic) or matching placebo, 1:1 allocation, for a period of 12 months. After 12 months, all participants in the placebo group will be crossed-over to receive Allo for the remainder of the study (6 month open-label phase). Brain imaging to evaluate the primary endpoint will be conducted at baseline, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women
* Age 55 to 80 years old
* Meets NIA-AA criteria for probable AD dementia
* MMSE of 20-26
* APOE ε4 positive
* Geriatric Depression Scale short form (GDS-S) score of ≤ 6
* No medical contraindications to participation
* Capacity to provide informed consent at screening

Exclusion Criteria:

* Dementia other than probable AD
* Use of benzodiazepines, anticonvulsants, antipsychotics, or other drugs that might interact with the GABA-A receptor complex
* History of stroke with a modified Hachinski Ischemic Scale score >4
* History of seizure disorder, focal brain lesion, traumatic brain injury
* History within the last 5 years of a primary or recurrent malignant disease
* Unstable or clinically significant cardiovascular, kidney or liver disease
* MRI indicative of any other significant abnormality, including but not limited to one or more significant ARIA-E or macro-hemorrhage findings, or multiple microhemorrhages (>8), or Fazekas score of 3; encephalomalacia, aneurysms, vascular malformations, subdural hematoma, or space occupying lesions
* Any conditions that would contraindicate MRI studies.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Hippocampal volume | Baseline to 12 months
  mm3

SECONDARY OUTCOMES:
Cambridge Cognition's Paired Associates Learning Test | Baseline to 12 months
  Total errors score (adjusted) - number of errors made by the participant (range: 0 to ~120). Higher scores indicate poor performance.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline to 12 months
  Composite score (higher score indicate better outcome)
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) 11 | Baseline to 12 months
  Total score (range 0 to 70); higher scores indicate poor performance.
Alzheimer's Disease Cooperative Study (ADCS) Instrumental Activities of Daily (iADL) Living (iADL) | Baseline to 12 months
  iADL subscore (range 0-56): Lower score indicates greater severity
Safety and tolerability | Baseline to 12 months
  Frequency of adverse events and serious adverse events

OTHER OUTCOMES:
Other regional brain volumes | Baseline to 12 and 18 months
  Change in regional brain volumes (mm3)
Diffusion tensor imaging (DTI) | Baseline to 12 and 18 months
  Change in white matter tract diffusion (scalar values and/or mm2/sec)
Resting state functional MRI | Baseline to 12 and 18 months
  Change in functional connectivity (z transformed correlations)
Arterial spin labeling (ASL) | Baseline to 12 and 18 months
  Change in regional cerebral blood flow (mL/100g)
Exploratory blood based biomarkers | Baseline to 12 and 18 months
  Change from baseline in biomarkers of AD pathology, neurogenesis and inflammation
Clinical Dementia Rating (CDR) | Baseline to 12 and 18 months
  Sum of boxes score (CDR-SB): range 0-18
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) 14 | Baseline to 12 and 18 months
  Total score (range 0-90)
Mini Mental State Examination (MMSE) | Baseline to 12 and 18 months
  Total score (range 0-30)
Neuropsychiatric Inventory-Questionnaire (NPI-Q) | Baseline to 12 and 18 months
  Total score (range 0-36). Higher scores indicate greater symptom severity
EuroQol 5-Dimension / 5-Level health-related quality of life scale scores (EQ-5D-5L) | Baseline to 12 and 18 months
  Reported as frequency, percentage and index value.
Quality of Life in Alzheimer's Disease scale (QoL-AD) | Baseline to 12 and 18 months
  Total score (range 13-52). Higher score indicate better QoL
Zarit Burden Interview (ZBI) | Baseline to 12 and 18 months
  Total score (range 0-48). Higher scores indicate high burden

CONTACTS AND LOCATIONS:
Overall Officials: Roberta D Brinton, PhD, Principal Investigator — University of Arizona; Lon Schneider, MD, Principal Investigator — University of Southern California; Gerson D Hernandez, MD, MPH, Study Director — University of Arizona
Locations (8):
- United States (8):
  - Perseverance Research Center, Scottsdale, Arizona
  - ATP Clinical Research, Costa Mesa, California
  - Syrentis Clinical Research, Santa Ana, California
  - Optimus U Corporation, Miami, Florida
  - Miami Jewish Health, Miami, Florida
  - Combined Research, Orlando, Florida
  - Conquest Research, Winter Park, Florida
  - MedVadis Research, Waltham, Massachusetts

REFERENCES:
- [Background] Raikes AC, Hernandez GD, Matthews DC, Lukic AS, Law M, Shi Y, Schneider LS, Brinton RD. Exploratory imaging outcomes of a phase 1b/2a clinical trial of allopregnanolone as a regenerative therapeutic for Alzheimer's disease: Structural effects and functional connectivity outcomes. Alzheimers Dement (N Y). 2022 Mar 14;8(1):e12258. doi: 10.1002/trc2.12258. eCollection 2022. PMID 35310526
- [Background] Hernandez GD, Solinsky CM, Mack WJ, Kono N, Rodgers KE, Wu CY, Mollo AR, Lopez CM, Pawluczyk S, Bauer G, Matthews D, Shi Y, Law M, Rogawski MA, Schneider LS, Brinton RD. Safety, tolerability, and pharmacokinetics of allopregnanolone as a regenerative therapeutic for Alzheimer's disease: A single and multiple ascending dose phase 1b/2a clinical trial. Alzheimers Dement (N Y). 2020 Dec 16;6(1):e12107. doi: 10.1002/trc2.12107. eCollection 2020. PMID 33344752
- [Background] Brinton RD. Neurosteroids as regenerative agents in the brain: therapeutic implications. Nat Rev Endocrinol. 2013 Apr;9(4):241-50. doi: 10.1038/nrendo.2013.31. Epub 2013 Feb 26. PMID 23438839
- [Background] Brinton RD, Wang JM. Therapeutic potential of neurogenesis for prevention and recovery from Alzheimer's disease: allopregnanolone as a proof of concept neurogenic agent. Curr Alzheimer Res. 2006 Jul;3(3):185-90. doi: 10.2174/156720506777632817. PMID 16842093